CLINICAL TRIAL: NCT02506556
Title: A Phase II Exploratory, Open-label, Single Arm Study of BYL719 Monotherapy, a Selective Phosphatidylinositol 3-kinase (PI3K) Alpha Inhibitor, in Adult Patients With Advanced Breast Cancer Progressing After First Line Therapy.
Brief Title: Phosphatidylinositol 3-kinase (PI3K) Alpha iNhibition In Advanced Breast Cancer
Acronym: PIKNIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LL14/02
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Last update posted 2022-08-16 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Breast Cancer
Keywords: Pi3K pathway
MeSH Terms: conditions — Breast Neoplasms | interventions — Alpelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- experimental (Experimental): BYL719 350 mg orally daily until progression, undue adverse events or withdrawal of consent.
  Interventions: Drug: BYl719

INTERVENTIONS:
Drug: BYl719 — Treatment: BYL719 350mg orally daily Treatment will be given daily until progression, undue adverse events or withdrawal of consent.
  Dose reductions (two levels) are allowed. Each cycle is 28 days

SUMMARY:
This is a phase II, exploratory, open-label, single arm study of BYL719 monotherapy, a selective phosphatidylinositol 3-kinase (PI3K) alpha inhibitor, in adult patients with advanced metastatic breast cancer progressing after first line therapy. Patients with advanced hormone receptor positive tumors will be required to have an alteration of the PI3K pathway. Those patients with advanced triple negative breast cancers are genetically unselected for this study.

DETAILED DESCRIPTION:
The primary purpose of this study is to determine whether BYL719 is a safe and effective drug treatment for adult patients with advanced breast cancer who have progressed after first line therapy.

Who is it for? Patients may be eligible to join this study if over 18 years old, male or female, with advanced metastatic or locally recurring breast cancer which has progressed after first line therapy.

Study details All participants enrolled in this study will take the study drug, BYL719, which is a selective phosphatidylinositol 3-kinase (PI3K) alpha inhibitor. This will involve taking tablets daily.

Participants will attend regular follow-up visits for up to 2 years in order to evaluate objective response rate, clinical benefit rate, progression free survival, safety and tolerability of treatment. Regular scans and blood tests will be performed

There will be two cohorts of participants involved in this study - those with metastatic triple negative breast cancer (TNBC) and those with estrogen receptor positive and HER2 negative (ER+/HER2-) breast cancers with a genetic mutation in the PI3K pathway. Efficacy and safety of BYL719 in these patients and associations with genetic features will be evaluated in order to try to identify biomarkers of response in breast cancer.

Study medication will be continued until disease progression, unacceptable toxicity or requirement to start another anti-cancer medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for inclusion in this study have to meet all of the following criteria:
* Males and females of any menopausal status
* Patient has signed the Informed Consent Form (ICF) prior to any screening procedures being performed and is able to comply with protocol requirements
* Age ≥ 18 years old
* Eastern Cooperative Oncology Group (ECOG) 0-2 that the investigator believes is stable at the time of screening
* Patient has locally recurrent (incurable) or metastatic disease
* Patient is able to swallow and retain oral medication
* Known HER2 status (local lab) that is negative on IHC (IHC=0) and/or non-amplified.
* Known estrogen receptor (ER) and progesterone receptor (PR) status (local lab)
* Recent tumor tissue must be available from a metastatic or recurrent lesion for next generation sequencing targeted gene panel
* Patients with triple negative breast cancer (TNBC) disease (ER<1%, HER2-negative) should have documented progression on at least one line of prior systemic therapy in the metastatic setting or within 12 months of adjuvant therapy completion. There is no limit on previous therapies. There will be no molecular selection of these patients.
* Patients with ER-positive (ER≥1%, HER2-negative) disease should have documented progression on at least one line of prior systemic endocrine therapy in the metastatic setting. There is no limit on previous therapies. Prior everolimus is allowed.
* Patients are defined as "PI3K abnormal" if they have documented gene mutation in AKT1,2,3,ALK, EGFR, ERBB2,3,4, HRAS, INPP4B, KRAS, NRAS, PTEN, PIK3CA, PIK3R1, PIK3R3, PTEN or gene amplification in EGFR, PIK3CA, PIK3R1 or loss in PTEN and INPP4B as per a next generation targeted gene sequencing panel
* Measurable disease by RECIST v 1.1 criteria or non- measurable disease that is clinically evaluable (bone only disease allowed if evaluable)
* Patient has adequate bone marrow and organ function assessed within 72 hours prior to first dose:
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
* Platelets ≥ 100 x 10^9/L
* Hemoglobin (Hgb) ≥ 9.0 g/dL
* Serum creatinine ≤ 1.5 x ULN
* Total serum bilirubin ≤ 1.5 x ULN (in patients with known Gilbert's syndrome, a total bilirubin ≤ 3.0 x ULN with direct bilirubin ≤ 1.5 x ULN)
* AST and ALT ≤ 2.5 x ULN (alternatively < 5 x ULN if evidence of liver metastases)
* Fasting blood glucose ≤ 140mg/dL or ≤ 7.8 mmol/L

Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria:

* Patient has a primary central nervous system (CNS) tumor or CNS tumor involvement.
* However patients with metastatic CNS tumors may participate in this study if the patient is:
* Four weeks from prior therapy completion (including radiation and surgery) to starting study treatment
* Clinically stable with respect to the CNS tumor at the time of screening
* Not receiving steroid therapy
* Patient with diabetes mellitus (fasting glucose >120mg/dl or 6.7 mmol/L), or documented steroid-induced diabetes mellitus
* Patient has a history of another malignancy within 2 years prior to starting study treatment, except for cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix.
* Patient who has not recovered to grade 1 or better (except alopecia) from related side effects of any prior antineoplastic therapy
* Patient who has had systemic chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to study entry.
* Patient who has received radiotherapy ≤ 4 weeks prior to starting study drugs, with exception of palliative radiotherapy (≤ 2 weeks prior to starting study drugs), who has not recovered from side effects of such therapy to baseline or Grade ≤ 1 and/or from whom ≥ 30% of the bone marrow was irradiated. Target lesions should not have had previous irradiation unless have progressed post treatment.
* Patient who has undergone major surgery ≤ 4 weeks prior to starting study treatment or who has not recovered from side effects of such procedure.
* Patient has a clinically significant cardiac disease or impaired cardiac function, such as:
* Congestive heart failure (CHF) requiring treatment (New York Heart Association (NYHA) Grade ≥ 2), left ventricular ejection fraction (LVEF) < 50% as determined by multi-gated acquisition (MUGA) scan or echocardiogram (ECHO)
* History or current evidence of clinically significant cardiac arrhythmias, atrial fibrillation and/or conduction abnormality, e.g. congenital long QT syndrome, high-grade/complete AV-blockage
* Acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass graft (CABG), coronary angioplasty, or stenting), < 3 months prior to screening
* QT interval adjusted according to Fredericia (QTcF) > 480 msec on screening ECG.
* Patient who has any severe and/or uncontrolled medical conditions such as:
* Active or uncontrolled severe infection,
* Liver disease such as cirrhosis, decompensated liver disease, and chronic hepatitis (i.e. quantifiable hepatitis B HBV-DNA and/or positive HbsAg, quantifiable hepatitis C HCV-RNA)
* Known severely impaired lung function (spirometry and DLCO 50% or less of normal and O2 saturation 88% or less at rest on room air)
* Active, bleeding diathesis;
* Uncontrolled arterial hypertension defined by blood pressure > 140/100 mm Hg at rest (average of 3 consecutive readings 5 min apart)
* Chronic treatment with corticosteroids or other immunosuppressive agent
* Patient who is currently receiving medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (TdP) and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug treatment.
* Patient who has participated in a prior investigational study within 30 days prior to enrollment.
* Patient who is currently receiving treatment with drugs known to be moderate or strong inhibitors or inducers of cytochrome isoenzymes CYP34A or CYP2C8. The patient must have discontinued moderate and strong inducers of both enzymes for at least one week and must have discontinued strong and moderate inhibitors before the start of treatment. Switching to a different medication prior to start of treatment is allowed; Refer to Appendix 1
* Patient with impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral BYL719 (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Patient with known positive serology for human immunodeficiency virus (HIV).
* Patients who have received live attenuated vaccines within 1 week of start of study drug and during the study. Patient should also avoid close contact with others who have received live attenuated vaccines. Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines.
* Pregnant or nursing (lactating) woman, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test (> 5 mIU/mL).
* Patient who does not apply highly effective contraception during the study and through the duration as defined below after the final dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-09-07 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Response is assessed from date of study enrolment every 2 cycles for the first 24 weeks and every 12 weeks after that or as clinically indicated until documented date of progression, death from any cause whichever came first assessed up to 60 months
  The percentage of patients who achieve a complete or partial response as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.

SECONDARY OUTCOMES:
Clinical Benefit Rate | Response is assessed from date of study enrolment every 2 cycles for the first 24 weeks and every 12 weeks after that or as clinically indicated until documented date of progression, death from any cause whichever came first assessed up to 60 months.
  Defined as Complete or partial responses according to RECIST 1.1 criteria or stable disease for 6 months or greater
Progression free survival | Defined as the time from study entry until documented disease progression. Patients will be followed up for a maximum of 2 years.
  Defined as the time from study entry until documented disease progression
Safety and tolerability of BYL719 | Safety is assessed by incident of adverse events according to NCI Common Toxicity Criteria for Adverse Effects (CTCAE) version 4 though out the study from until documented one month post cessation of study medication - on average 8 months
  Safety and tolerability will be described using frequency of significant treatment related adverse events (AEs) using CTCAE 4.0 grade ≥3, all Serious Adverse Events and SUSARs. Safety analysis will include all patients who have received at least one dose of the drug and will be evaluated descriptively

CONTACTS AND LOCATIONS:
Overall Officials: Sherene Loi, MD,PhD, Study Chair — Peter MacCallum Cancer Centre, East Melbourne, Victoria, AUSTRALIA
Locations (1):
- Peter MacCallum Cancer Centre, East Melbourne, Victoria, Australia

REFERENCES:
- [Background] Zardavas D, Phillips WA, Loi S. PIK3CA mutations in breast cancer: reconciling findings from preclinical and clinical data. Breast Cancer Res. 2014 Jan 23;16(1):201. doi: 10.1186/bcr3605. PMID 25192370
- [Background] Loi S, Michiels S, Lambrechts D, Fumagalli D, Claes B, Kellokumpu-Lehtinen PL, Bono P, Kataja V, Piccart MJ, Joensuu H, Sotiriou C. Somatic mutation profiling and associations with prognosis and trastuzumab benefit in early breast cancer. J Natl Cancer Inst. 2013 Jul 3;105(13):960-7. doi: 10.1093/jnci/djt121. Epub 2013 Jun 5. PMID 23739063
- [Background] Loi S, Haibe-Kains B, Majjaj S, Lallemand F, Durbecq V, Larsimont D, Gonzalez-Angulo AM, Pusztai L, Symmans WF, Bardelli A, Ellis P, Tutt AN, Gillett CE, Hennessy BT, Mills GB, Phillips WA, Piccart MJ, Speed TP, McArthur GA, Sotiriou C. PIK3CA mutations associated with gene signature of low mTORC1 signaling and better outcomes in estrogen receptor-positive breast cancer. Proc Natl Acad Sci U S A. 2010 Jun 1;107(22):10208-13. doi: 10.1073/pnas.0907011107. Epub 2010 May 17. PMID 20479250